CLINICAL TRIAL: NCT00938782
Title: A Prospective, Randomized, Double-Blinded Study of the Effect on Improved Recovery Using the SEDLine TM for the Titration of Sevoflurane in Elderly Patients Undergoing Non-Cardiac Surgery After Beta-Adrenergic Blockade
Brief Title: Using the SEDLine for the Titration of Sevoflurane in Elderly Patients Recovery Using the SEDLine TM for the Titration of Sevoflurane in Elderly Patients Undergoing Non-Cardiac Surgery After Beta-Adrenergic Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, David R. Drover, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU-11062007-818
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Monitoring with SEDLine Monitor (Active Comparator): Patient group randomized to active monitoring with SEDLine monitor for titration of anesthesia.
  Interventions: Device: Sedline
- Blinded monitoring with SeEDLine Monitor (No Intervention): Patient group randomized to blinded monitoring with SEDLine monitor for titration of anesthesia. Data captured but not used for titration of anesthesia.

INTERVENTIONS:
Device: Sedline
  Arms: Active Monitoring with SEDLine Monitor

SUMMARY:
Asses the effect of the use of Patient State Index (PSI) monitoring on difference in emergence profiles in the elderly (age >65 yrs) population to develop a cost-benefit profile.

Assess differences in Quality of Life using the QoR-40 (a validated 40-item questionnaire on quality of recovery from anesthesia) between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female.
* Patient is 65 years of age or older.
* Patient has a physical status between ASA I and III. (Appendix C).
* Patient scheduled for general anesthesia for non-cardiac surgery expected to last at least one hour.
* Patient able to communicate in English.
* Patient has signed an approved informed consent.

Exclusion Criteria:

* Patient's age is less than 65 years
* Anesthetic duration of less than one hour expected
* Treatment of beta blockers contra-indicated
* Not a candidate for general anesthesia
* Patient requires regional anesthesia with general anesthesia.
* ASA physical status of IV or V. (Appendix C)
* Patient has known drug or alcohol abuse.
* Patient has scalp or skull abnormalities such as psoriasis, eczema, angioma, scar tissue, burr holes, cranial implants (such as plates, shunts, etc.).
* Patient has experienced a head injury with loss of consciousness within the last year.
* Patient has known neurological and psychiatric disorder that interferes with the patient's level of consciousness.
* Known concurrent chronic usage of psychoactive or anticonvulsive drugs within the last 90 days, or any use in the last 7 days (i.e. tricyclic antidepressants, MAO inhibitors, lithium, SSRIs, neuroleptics, anxiolytics or antipsychotics).
* Patient has any medical condition which, in the judgment of the investigator, renders them inappropriate for participation in this study, such as Guillen Bare syndrome
* Known hypersensitivity to the intended anesthetic agents including significant post-operative nausea or vomiting.
* Uncontrolled hypertension (unresponsive to medication): Systolic BP > 180 mmHg or Diastolic BP > 105 mmHg
* Pre-Op baseline heart rate < 45 beats per minute
* Weight 50% greater than ideal body weight
* Already monitored for EP or EEG, i.e., Spinal cord cases
* Actual anesthetic duration < 1 hour (assessed after emergence).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Drover, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Drover DR, Schmiesing C, Buchin AF, Ortega HR, Tanner JW, Atkins JH, Macario A. Titration of sevoflurane in elderly patients: blinded, randomized clinical trial, in non-cardiac surgery after beta-adrenergic blockade. J Clin Monit Comput. 2011 Jun;25(3):175-81. doi: 10.1007/s10877-011-9293-1. Epub 2011 Aug 10. PMID 21830049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Surgical patients older than 65 years of age receiving beta-adrenergic blockers for a minimum of 24 hours preoperatively were randomized to two groups.
Groups:
- 1 - SEDLine™ Group: Surgical patient group randomized to active monitoring with Sedline monitor plus other routine monitors. Anesthesia protocol developed with respect to titrate based on vital plus Sedline monitor.
- 2- Control Group: Surgical patient group randomized to active monitoring with Sedline monitor plus other routine monitors. Anesthesia protocol developed with respect to titrate based on physiologic vitals without input from Sedline monitor.
Period: Overall Study
Arm/Group | 1 - SEDLine™ Group | 2- Control Group
Started | 32 (Pre-induction of anesthesia) | 35 (Monitoring started pre-induction of anesthesia)
Completed | 32 (Upon discharge from PACU) | 35 (Upon discharge from PACU)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Surgical patients older than 65 years of age receiving beta-adrenergic blockers for a minimum of 24 hours preoperatively were randomized to two groups.
Groups:
- 1 - SEDLine™ Group: Surgical patient group randomized to active monitoring with Sedline monitor plus other routine monitors. Anesthesia protocol developed with respect to titrate based on vital plus Sedline monitor.
  Surgical patients older than 65 years of age receiving beta-adrenergic blockers for a minimum of 24 hours preoperatively were randomized to two groups: a group whose titration of sevoflurane was based on SEDLine™ data (SEDLine™ group).
- 2 - CONTROL Group: Surgical patient group randomized to active monitoring with Sedline monitor plus other routine monitors. Anesthesia protocol developed with respect to titrate based on physiologic vitals without input from Sedline monitor.
  Surgical patients older than 65 years of age receiving beta-adrenergic blockers for a minimum of 24 hours preoperatively were randomized to two groups: a group whose titration of sevoflurane was not based on SEDLine™ data (CONTROL group)
- Total: Total of all reporting groups
Arm/Group | 1 - SEDLine™ Group | 2 - CONTROL Group | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (5.7) | 74.5 (6.7) | 74.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 20 | 24 | 44
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation
Description: The exact time from end of last anesthetic drug to time of tracheal extubation.
Time Frame: Measured from time of end anesthesia to time of tracheal extubation.
Population: All patients enrolled in both groups.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 1 - Sedline Group: Patient group randomized to active monitoring with Sedline monitor.
- 2 - Control Group: Patient groups randomized to active monitoring versus blinded monitoring. This group had teh clinician blinded to output of the Sedline monitor.
Arm/Group | 1 - Sedline Group | 2 - Control Group
Number analyzed (Participants) | 32 | 35
minutes | 13.0 (5.9) | 12.5 (7.4)

ADVERSE EVENTS:
Time Frame: 1 day during anesthesia period
Groups:
- 1 - SEDLine Group: Patient groups randomized to active monitoring. This group had Sedline monitor used to titrate anesthesia.
- Group 2 - Control Group: Patient groups randomized to monitoring with blinded data not used to titrate anesthesia.
Arm/Group | 1 - SEDLine Group | Group 2 - Control Group
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No